CLINICAL TRIAL: NCT00005948
Title: A Pilot Study of High Dose Busulfan Combined With IL2/GM-CSF Activated Autologous/Syngeneic PBSC, Sequential IL2/GM-CSF Therapy and Alpha Interferon Maintenance Therapy as Treatment of CML
Brief Title: Chemotherapy Followed by Peripheral Stem Cell Transplantation And Biological Therapy in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1455.00; FHCRC-1455.00; NCI-G00-1792; CDR0000067877 (Registry Identifier: PDQ)
Record Dates: First submitted 2000-07-05; First posted 2004-04-02 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Leukemia
Keywords: relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase | interventions — aldesleukin; Interferon-alpha; sargramostim; Busulfan; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant interferon alfa
Biological: sargramostim
Drug: busulfan
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy followed by peripheral stem cell transplantation and biological therapy in treating patients who have chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity of high-dose busulfan followed by interleukin-2 (IL-2) and sargramostim (GM-CSF) activated autologous/syngeneic peripheral blood stem cell (PBSC) transplantation, sequential IL-2 and GM-CSF therapy, and interferon alfa in patients with chronic myelogenous leukemia. II. Determine engraftment potential of IL-2/GM-CSF activated PBSC followed by sequential IL-2/GM-CSF therapy in this patient population. III. Assess the time to cytogenetic and/or morphologic relapse, overall event-free survival, and overall survival in these patients treated with this regimen.

OUTLINE: Autologous peripheral blood stem cells (PBSC) are harvested and activated with interleukin-2 (IL-2) and sargramostim (GM-CSF) on another protocol. Patients receive oral busulfan every 6 hours on days -6 to -3 for a total of 16 doses. IL-2 and GM-CSF-activated PBSC are reinfused on day 0. Beginning 4 hours after PBSC infusion, patients receive IL-2 IV continuously for 5 days followed by 2 days of rest for 4 weeks. In addition, GM-CSF is administered subcutaneously (SC) every Monday, Wednesday, and Friday for 4 weeks. Upon hematologic recovery, but no earlier than 2 weeks after IL-2 and GM-CSF, patients receive interferon alfa SC 3 times weekly until clear evidence of disease progression. Patients are followed every 6 months for 3 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Chronic myelogenous leukemia with previously stored CD34 cells from FHCRC-928.00 Chronic phase: No evidence of a major response after 6-month course of interferon alfa OR Initially achieved a major cytogenetic response but subsequently failed interferon alfa OR Accelerated phase: At least 1 month after collection of peripheral blood stem cells No blast crisis No CNS involvement Ineligible for or refused allogeneic conventional or minitransplant protocol

PATIENT CHARACTERISTICS: Age: 70 and under Performance status: Karnofsky 80-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL (unless history of Gilbert's disease) AST or ALT no greater than 2.5 times upper limit of normal No cirrhosis Hepatitis B and C negative Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No myocardial infarction within past 12 months No unstable angina, poorly controlled arrhythmias, or hypertension LVEF greater than 50% Pulmonary: DLCO at least 50% Alveolar arterial gradient less than 30 at sea level Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception HIV negative No active infection requiring systemic antibiotics No known allergy to gentamicin or murine or E. coli proteins or documented prior anaphylactic reaction to sargramostim (GM-CSF) or interleukin-2

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: Not specified Endocrine therapy: No concurrent ongoing steroids Radiotherapy: Not specified Surgery: Not specified

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-01; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona A. Holmberg, MD, PhD, Study Chair — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - University of Colorado Cancer Center, Denver, Colorado
  - Fred Hutchinson Cancer Research Center, Seattle, Washington